CLINICAL TRIAL: NCT02870439
Title: Testing an Innovative Biomarker: Expression of HIF-1α and Its Isoforms in the Blood and Skin Tissue of Major Burns
Acronym: HIF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-23; 2012-A00786-37 (Other: Ansm)
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Burn Injuries
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- patients with at least 20% of wounded burns body (Experimental)
  Interventions: Other: Blood drawn
- patients with at least 5% of wounded burns body (Experimental)
  Interventions: Other: Blood drawn
- patients with post-surgical wounds with skin resection (Experimental)
  Interventions: Other: Blood drawn

INTERVENTIONS:
Other: Blood drawn

SUMMARY:
Burn injury with full-thickness skin damage that encompass large body surface areas can induce local and systemic perturbations that are costly in terms of human suffering as well as in strains on the health care system. Characterization of new major molecular biomarkers involved in this process creates significant diagnostic and therapeutic challenges.

Hypoxia-inducible factor-1 α (HIF-1 α) is a ubiquitously expressed heterodimeric transcription factor comprising an α and a β subunit. It was shown that under normoxic conditions, the HIF-1α subunit is ubiquitinated and degraded, whereas under hypoxic conditions, HIF-1α accumulates, dimerizes with HIF-1β, and activates the transcription of a spectrum of target genes encoding multiple angiogenic growth factors and cytokines of potential importance in wound healing. Seven isoforms of HIF-1α issued from alternative splicing have been identified.

The importance of HIF-1α in wound healing in animal models has been suggested by several studies. Indeed, diminished HIF-1 levels and activity have been documented in conditions of impaired wound healing. The literature review shows a marked reduction of HIF-1α levels in mice in case of burn wound skin that in the case of excisional cutaneous wound. Other studies have shown that the expression of HIF-1α was correlated with the extent and depth of the burns.

This study aims to improve the knowledge on the pathophysiological factors involved in the field of wound healing. The assumptions are based on results of studies done on mice, and this work aims to document these findings in humans.

Objective

The main objective of the study is to compare the variations of expression of HIF-1α measured in blood and skin tissue samples in three groups:

* Subjects with major burn wounds involving more than 20% of the total body surface area;
* Subjects with burn wounds smaller than 5% of total body surface area;
* Subjects with a skin wound after a surgical procedure requiring a skin resection.

Secondary objectives are to compare the expression levels of HIF-1α locally at the burn site to those observed in blood, to evaluate the expression of growth factors produced by HIF-1α target genes (VEGF and EPO) or playing a central role in the healing process (TGF-β1), and to assess the correlation between the expression of HIF-1α and the kinetics of wound healing of the subject rated by evaluation of time of donor sites complete epithelialization.

Material and Methods

We propose to create three groups:

* 15 patients with extensive third degree burns involving more than 20% of the total body surface area;
* 15 patients with less extensive third degree burns, involving less than 5% of body surface area;
* 15 patients with post-surgical wounds with skin resection. Skin and tissue specimens will be collected three times: day 0, 7 and 14 from burned patients (with more than 20% of the total body surface area and less than 5% of body surface area). Samples of skin tissue will be collected within the skin resection from patients with post-surgical wounds at day 0, blood samples will be collected at day 0 and 14.

ELIGIBILITY:
Inclusion Criteria:

* Patient with burn wounds

Exclusion Criteria:

* Patient with wounds coming from electrical or chemical burns
* Patient undergoing long term corticotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
percentage of the variations of expression of HIF-1α | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille; Aurélie HAUTIER, MD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No